CLINICAL TRIAL: NCT03656237
Title: The Impact of Case-based Focused Low-dose High-frequency hands-on Training of Facility Health Care Providers and Community Health Workers on Maternal and Newborn Health in Mali, a Cluster Randomized Trial.
Brief Title: Low-dose High-frequency Training of Facility Health Care Providers in Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Red Cross (Other); Global Affairs Canada (Other); Croix Rouge Malienne (Unknown); University of the Sciences, Techniques and Technologies of Bamako (Other); Direction Nationale de la Santé Mali (Unknown)
Responsible Party: Principal Investigator, Diego Bassani, Director, International Program Evaluation Unit (IPE), Center for Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1000060635
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Perinatal Mortality
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial (Clusters are the community health units - CSCOMs)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual training + Audits + LDHF training (Experimental): Usual training of health workers, in classroom, following standard curriculum
  + Mortality and Morbidity Audits in facility every two weeks followed by LDHF training focused on gaps in knowledge or practice identified during the audits
  Interventions: Other: Usual Training; Other: Audits + LDHF Training
- Audits + LDHF training (Experimental): Mortality and Morbidity Audits in facility every two weeks followed by LDHF training focused on gaps in knowledge or practice identified during the audits
  Interventions: Other: Audits + LDHF Training
- Usual Training (Active Comparator): Control Arm exposed to usual training of health workers, in classroom, following standard curriculum
  Interventions: Other: Usual Training

INTERVENTIONS:
Other: Usual Training — Training in a classroom setting of health care providers
  Other Names: Classroom Training
  Arms: Usual Training; Usual training + Audits + LDHF training
Other: Audits + LDHF Training — Clinical audits followed by case-based low-dose high-frequency training
  Other Names: Mort. Morb. Audit + Low-dose High-freq. training
  Arms: Audits + LDHF training; Usual training + Audits + LDHF training

SUMMARY:
This 3-arm cluster randomized trial (C-RCT) has the following objectives:

Primary Aim

To evaluate the effectiveness of an on-site case-based focused low-dose high-frequency training strategy in a primary health care facility labour room, during the provision of care to mothers and newborns, through childbirth and within seven days post-partum for the healthcare providers and the community health workers linked to the health facility in decreasing perinatal mortality.

Secondary Aims

To determine if introduction of an on-site case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting reduces:

* Perinatal morbidity incidence
* Post-partum Hemorrhage

To determine if introduction of an on-site case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting increases ENC practices:

* Early initiation and exclusive breast feeding
* Thermal protection (prevention of hypothermia)
* Clean cord care
* Delayed bathing
* Resuscitation-Initiation of breathing

To determine if introduction of a case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting for CHWs decreases:

* Delayed Identification of danger signs during pregnancy, labour and perinatal period
* Delayed referral of complicated cases during pregnancy, labour and perinatal period

To determine the cost effectiveness of a case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting

DETAILED DESCRIPTION:
Hypothesis The investigators hypothesize that on-site case-based focused low-dose high-frequency hands on training of maternal and neonatal health care providers and community health workers will have an impact on reducing perinatal mortality rate (PMR) in comparison to Maternal Newborn and Child Health (MNCH) refresher training in a classroom setting.

Primary Aim To evaluate the effectiveness of an on-site case-based focused low-dose high-frequency training strategy in a primary health care facility labour room, during the provision of care to mothers and newborns, through childbirth and within seven days post-partum for the healthcare providers and the community health workers linked to the health facility in decreasing perinatal mortality.

Secondary Aims

To determine if introduction of an on-site case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting reduces:

* Perinatal morbidity incidence
* Post-partum Hemorrhage

To determine if introduction of an on-site case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting increases Early Newborn Care (ENC) practices:

* Early initiation and exclusive breast feeding
* Thermal protection (prevention of hypothermia)
* Clean cord care
* Delayed bathing
* Resuscitation-Initiation of breathing

To determine if introduction of a case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting for Community Health Workers (CHW) decreases:

* Delayed Identification of danger signs during pregnancy, labour and perinatal period
* Delayed referral of complicated cases during pregnancy, labour and perinatal period

To determine the cost effectiveness of a case-based focused low-dose high-frequency training methodology in comparison to MNCH refresher training in a classroom setting

Methodology

The study is designed as a facility based, cluster randomized, pragmatic, intervention trial. It will be conducted within the country's existing health care system. Specifically, the intervention is a comparison between 3 training modalities; (i) MNCH refresher training in a classroom setting (Ministry of Health (MoH) Mali) and clinical audits followed by on-site case-based focused low-dose high-frequency training of health care providers, (ii) clinical audits followed by on-site case-based focused low-dose high-frequency training of health care providers and (iii) a control group receiving only the MNCH refresher training in a classroom setting (MoH Mali) of health care providers. The standard MNCH refresher training will be delivered by government trainers as per Canadian Red Cross (CRC) planned program in Koulikoro region and the on-site case-based focused low-dose high-frequency trainings will be delivered by MoH trained trainers employed by SickKids and retrained on case-based focused low-dose high-frequency trainings and clinical audits (Figure I: C-RCT Flow Chart). Analysis will be intention to treat (ITT), taking into account the clustering of observations.

Randomization

Cluster Definition

A cluster is defined as the population residing in the catchment area of the primary health care facility (CSCom) and the stratification will be at the CSCom level. The primary health care facility (CSCom) provides basic maternal and newborn care services; catering to a population group (5000-10000) residing within a 10-15 Km radius. A community health worker is assigned to 1500 people (approximately 250 households) dispersed across up to 3 villages and provides services in areas 5Km or more away from a CSCom.

Randomization of clusters will be performed by an epidemiologist not directly involved in the research project and who is therefore unbiased regarding the randomization. Due to the nature of the intervention, blinding is not possible, however to ensure reduced measurement bias, data on the effect of the intervention will be collected by independent data collectors not involved in the intervention delivery. Randomization will be performed at the health facility level (primary health care facility-CSCom, catering to a population group of 5000-10000, residing within a 10-15 Km radius).

Study Setting The study will be conducted in four districts- Koulikoro, Kolokani, Banamba and Dioïla of Koulikoro Region, Mali, within the CRC MNCH program area with a 4-year timeline: 2016-2020. Koulikoro region was chosen because of high perinatal mortality and morbidity indicators; however, these districts were also chosen for study logistics and administrative reasons; Mali Red Cross has a strong presence here due to projects involving strengthening of: CHWs and volunteers for MNCH related activities at iCCM sites. Political stability and availability of population and health facility assessment data from a CRC program baseline survey in 2016 were also taken into account.

Koulikoro Region is the second-most-western region of Mali. It covers an area of 90,120 square kilometers with an estimated 2009 population of 2,418,305 and a density of 26.83 people per square kilometers of land area. Mali's estimated birth rate is 42.91 per 1000 population (World Bank 2015) and the region of Koulikoro has an estimated perinatal mortality rate of 30 per 1000 live births with 49 % of births taking place at the CSCom level (CRC HHS 2016). Koulikoro region is separated in seven cercles: Kati, Kangaba, Koulikoro, Kolokani, Nara, Banamba and Dioïla. CRC/MRC program area encompasses the latter five. Of these, four districts (Koulikoro, Kolokani, Banamba and Dioïla) will be included in this study (Figure II: RCT Districts Profile).

Field operations for the study will be managed and coordinated by Dr. Moctar Tounkara, L'Université des Sciences, des Techniques et des Technologies de Bamako (USTTB), Mali.

Phase I: Study Duration The first phase of the study will be 6 months in total (July-December 2018) during which on-site case-based focused low-dose high-frequency trainings will be undertaken in 56 CSComs (Intervention Arm I and II). All facility births and any newborn referred to the health facility within 7 days of birth (irrespective of the place of birth) during phase I will be included in the final analyses. Data collection during this phase will commence two weeks after the first round of clinical audits and on-site case-based focused low-dose high-frequency trainings. Simultaneous data collection will occur in the 28 control CSComs. The timeline of the study can be seen in Figure IV: Timeline of the Trial.

Phase II: Study Duration The second phase of the study, which will focus on the collection of mortality and morbidity data (see section 16 for further details), will begin in January 2019 and extend for a total of 12 months. Therefore, approximately 17-18 months of births (30,000 newborns, based on 2016 CSCom births) will be included in the final analysis (Phase I and II combined). There will be a 3 month period to analyse the data and prepare the final report (Jan-March 2020). The timeline of the study can be seen in Figure IV: Timeline of the Trial.

Eligibility Criteria and Enrolment Study Population Eligibility All CSComs within participating clusters (CRC program area) with facility deliveries, perinatal referrals and affiliated community health workers will be eligible for enrollment in this study.

Enrolment

* Approval from the Ministry of Health Mali and the Regional Directorate of health, Koulikoro will be obtained to enroll CSComs in target districts providing basic obstetric and neonatal care and affiliated CHWs in the study.
* Key personnel from Regional Directorate of health, Koulikoro, will be oriented on the proposed operational research intervention.
* Subsequently the study team members will visit all eligible CSComs and share the letters of approval from the MoH and regional directorate with the facility in-charge to formalize the enrollment.
* All consenting women delivering a baby in the health facility will be enrolled in the study.
* All facility births and newborns referred to a health facility within the perinatal period with consenting parents will be enrolled in the study.

Intervention Arms Pre-Intervention Training (part of CRC/MRC project) Two maternal and neonatal health care providers from each CSCom in the Intervention Arm I will receive the MNCH refresher training in a classroom setting on AMTSL, ENC and PNC. The CHWs in Intervention Arm I and II will receive the MoH Mali iCCM and health education trainings in a classroom setting.

Intervention Arm I- Clinical audits and on-site case-based focused low-dose high-frequency trainings (detailed below).

Arm II- Clinical audits and on-site case-based focused low-dose high-frequency trainings (detailed below) Case-based focused low-dose high-frequency Training of HCPs and CHWs The intervention is a cluster level on-site case-based focused low-dose high-frequency training strategy offered to health facility staff providing basic obstetric and neonatal care and to community health workers providing maternal, neonatal health education, identification of danger signs for pregnant females during pregnancy and labour, newborns during delivery (home deliveries) and perinatal period, stabilization and timely referral.

Clinical Audits

In Mali, it is currently mandatory to notify maternal, perinatal and neonatal deaths/adverse events within 48 hours through the Integrated Disease Surveillance and Response Network; and to convene an audit of the same within 15 days of notification. These audits are being implemented throughout the country by the MOH and; will serve as the platform for the identification of cases for the case-based focused low-dose high-frequency trainings.

An audit committee comprising of health facility manager, basic obstetric and neonatal care providers and district/regional Health department representative will be formed (as per MoH Mali Guidelines-Annex I). An audit meeting will be convened bi-weekly facilitated by the intervention trainer.

All audit case summaries will be discussed in detail, identifying causes of death, complications and assessing the quality of care provided. The findings will be evaluated against existing service delivery standards/protocols. The clinical audit will identify knowledge deficit among health care providers, knowledge-to-action gap, and training requirements.

A biweekly mortality audit calendar will be developed for the 56 intervention CSComs (12 audits per CSCom over 6 months). For the intervention arms, MoH trainers, trained on the implementation of the intervention, will participate in the audits, facilitate the process and identify key areas for on-site case-based focused low-dose high-frequency training, mentoring and supervision of MNCH care providers.

A health facility representative designated by the audit committee will be responsible for providing audit support that includes providing medical records and supporting documentation to audit committee (Annex II), assisting in the development of process, procedural walk-throughs, and responding to various inquiries to assist the committee with the development and documentation of their work papers. Data from the patient's hospital record and CSCom DHIS2 will be used to compile mortality and morbidity audit documents and each case to be audited will be anonymized (Date, Time Patient and HCP identities), and summarized by the health facility representative nominated by the audit committee.

Factors external to the CSCom services which adversely affected patient outcome (such as delayed recognition of danger signs during pregnancy/labour with delayed referral, delayed recognition of danger signs during perinatal period with delayed referral) will be identified during the audit. These gaps will be addressed through case-based trainings of the community health workers at the corresponding CSCom.

The summary of each audited case will have a section to document action points for proposed trainings and managerial support, the same will also be recorded in the minutes of the audit committee meeting.

Following the audit committee meeting, the intervention trainer will stay on at the health facility for one more consecutive day to implement case-based focused low-dose high-frequency trainings to the CSCom staff providing basic obstetric and neonatal care and to community health workers linked to each CSCom.

This intervention will align with the existing MoH Mali program and not change the existing schedule of service delivery and training curricula (AMTSL, ENC, PNC, MoH-CHW Training) at the CSCom or for the CHWs. This approach will facilitate later scale-up of the proposed training strategy within the existing program in other districts of Koulikoro.

Control Arm:

As per MOH-Mali, directive clinical audits are to be implemented in all health facilities in the Koulikoro region, but there will be no on-site case-based focused low-dose high-frequency trainings resulting from the findings of these audits in the control arm during study duration. The CSCom staff and CHWs in the control area will only receive the MNCH refresher multi-method classroom trainings planned as part of CRC/MRC project. Two maternal and neonatal health care providers from each CSCom in the control arm will be trained on AMTSL, ENC, PNC, and the CHWs in iCCM and health education.

Health Facility and CHW Statistical Record All health facility staff and CHW's in the intervention and control arms will receive training on data collection and recording, in an effort to improve HMIS data quality, as part of the CRC/MRC planned program in Koulikoro region. HCP's and CHW's in both the intervention and control sites will receive this training prior to the initiation of the study.

Study Trainers:

Intervention trainers (11) will be selected according to the following criteria:

1. Obstetrician, Gynecologist or a General Duty Physician experienced in Obstetrics
2. Preferably resident of the intervention district
3. Previous experience with mortality audit process would be preferred

Intervention trainers will be trained on case-based focused low-dose high-frequency training strategy for Active Management of Third Stage of Labour (AMTSL), Essential Newborn Care (ENC), Postnatal Care (PNC), identification of danger signs for pregnant females during pregnancy and labour, newborns during delivery (Health facility and home deliveries) and perinatal period, stabilization, timely referral and facilitating maternal and perinatal mortality/morbidity audits by Master Trainers (MoH Mali/SK).

After completion of training, the trainers will visit assigned CSComs and conduct:

1. An introductory orientation meeting with the facility staff and CHWs on the proposed trial for approximately an hour.
2. A 2 day training on the processes of team building, and clinical audit for an interdisciplinary team comprising of the health facility manager, maternal and neonatal health care providers.

Implementation of maternal and perinatal mortality and morbidity audit at the CSComs will commence two weeks after this initial visit.

Logistics Data collectors Independent local data collectors (10) having completed secondary education will be hired and will undergo 5 days of formal training (5 data collectors will cover 8 CSComs and 5 will cover 9 CSComs each). As part of this training, data collectors will gain an in-depth understanding of all data collection forms and verbal autopsy process. Data collectors will conduct observed interactions (respondent interview) with a real mother having a live newborn as part of their training.

Data Collection Informed consent will be taken from all participants in the study and it will be made clear that eligible participants are under no obligation to participate in this study. In addition, the time burden associated with being involved in this study will be clearly outlined during the consent process.

A record of implementation and frequency of clinical audits conducted will be maintained in intervention arms I, II and control arm for the complete duration of this study- July 2018-December 2019.

i) Data collectors will visit CSComs in the intervention and control clusters once a month and after taking consent from the facility manager will collect data from the health facility record (labour room register, maternity ward register, DHIS2) for all deliveries pertaining to PPH, maternal deaths, still births, perinatal deaths, and complications related to labour and delivery for both the mother and newborn since her/his last visit. The data collector will also create a list of facility stillbirths and perinatal deaths with names and addresses for subsequent verbal autopsies (VA) after the 40-day bereavement period.

ii) In case of a still birth or neonatal death; an adult (husband/relative) will be tactfully requested to propose a convenient time and venue for the respondent interview that will be conducted by a data collector. The parents/relatives will be given the choice of whether or not a verbal autopsy can be performed around the events surrounding the stillbirth or death of the newborn (VA occurs 40 days after the death). Further details on the verbal autopsy are included in section 20.

iii) The data collector will also conduct a follow-up home visit for all CSCom births and referrals in her/his catchment area and administer a short questionnaire (Questionnaire Form II-Annex IV) after taking consent from the parent/caregiver of the newborn after day 8 post-birth to capture any complications/adverse events and current status of the newborn. If the mother or caregiver is unavailable at the time of the home visit, the visit will be rescheduled to the earliest available time. If the newborn is not alive, the data collector will leave after recording the date, time and if possible the probable cause of death and return after the 40 day bereavement period to conduct a verbal autopsy. Further details on the verbal autopsy are included in section 20.

For newborns who do not complete their study visit on or after day 8 post-birth, all available data from the health facility record will be collected in order to ascertain the maternal and perinatal outcome (mortality and morbidity during perinatal period).

iv) The parents of a newborn who was not delivered in the CSCom but was referred to it within 7 days of birth will be administered the household questionnaire by the data collector on or after day 8 of life.

The intervention trainer will collect audit attendance and content data (Annex VI):

1. Audit date, time, participants and their roles
2. List of issues discussed and training needs identified
3. Summary of trainings conducted with dates following the audit
4. List of trainees (HCP/designation and CHWs)

   19) Field Supervision and Quality Control An In-country project team composed of a study manager and coordinator with the help of 4 field-monitoring officers will coordinate project activities. . The project team will also be responsible for all the logistics and monitoring support of project activities in addition to oversight.

   Field supervisors will be responsible for ensuring quality control in data collection as well as maintain close liaison with the CSComs and communities. They will also be responsible to randomly back check the CSCom and field data as part of quality control in data collection. They will also ensure timely and accurate electronic data transfer from field to the study coordinator. The study manager will have overall responsibility for the on-ground management and supervision of the trial.

   Data Safety Monitoring A data and safety monitoring board (DSMB) will be convened with three individuals, Dr. Lisa Pell, The Hospital for Sick Children, Professor Ibrahim TEGUETE, Obstetrician Gynecologist, USTT, Mali and, Professor Mariam SYLLA pediatrician, USTT, Mali with expertise in the clinical area of the trial. The DSMB will have the mandate of making an independent, fully informed assessment of the progress of the trial. It will make recommendations to the trial PI as to whether to continue, amend or terminate the trial. The DSMB will be provided de-identified data at 6th and 12th month of data collection. The identity of study groups will be masked unless the DSMB determines that the identities of the groups are necessary for their decision making. The DSMB may also make recommendations / escalate issues to the REB at SickKids (primary organization) and Comité d'éthique de la Faculté de Médecine, de Pharmacie et d'Odonto-Stomatologie de Mali (FMPOS).

   The investigators will adopt a stopping rule for harm (higher than probability of higher mortality in the intervention arm) based on Bayesian probabilities estimated during interim analysis at the following times (t) mid-point (8 months) and again at 12 months of trial duration (post intervention rollout (+0.5 months). The investigators will use a skeptical prior for the Bayesian analysis, a distribution that attempts to formalize the belief that treatments are unlikely to be different. The trial is going to be stopped at time t if D(t) is at least equal to 95 percent. D(t) is the predictive probability that the survival function in the intervention group is smaller than the survival function in the placebo group at time t.

   Function / Responsibilities of the DSMB:
   * Assess and monitor the trial from an ethical perspective
   * Assess the quality and completeness of interim data
   * Review recruitment and participant retention data
   * Review protocol and deviations from the Standard Operating Procedures
   * Review any individual events considered significant
   * Make recommendations regarding trial continuation, amendments or termination
   * Assess the need for stopping the trial prematurely based on strong evidence of unintended harm or external evidence for all or any of the following:

     1. Failure to adhere to the research protocol and non-compliance with goals for recruitment and retention.
     2. Any factors that might affect the study outcome or compromise the confidentiality of the trial data (such as protocol violations, unmasking, etc.); and, c) Factors external to the study such as scientific or therapeutic developments that may impact participant safety or the ethics of the study.

   Ethical Approval, Consent Process, Confidentiality, and Safety Ethical Approval The study proposal will be submitted for ethical approval to Comité d'éthique de la Faculté de Médecine, de Pharmacie et d'Odonto-Stomatologie de Mali (FMPOS), and the Research Ethics Board at The Hospital for Sick Children, Toronto, Canada. Subsequent to this approval, consent and agreement to participate will be obtained from the regional and district health departments of Koulikoro, Kolokani, Banamba and Dioïla in Koulikoro, Mali.

   Participant Consent Written consent will be obtained from mothers and/or fathers of newborns at the follow-up household visit and also for verbal autopsy. If the mother is not able to give consent, her husband or other adult family member present will be requested to give consent to participate in the study. If the respondent cannot read, the consent statement will be read to her/him and a thumb impression by the respondent in place of a signature will signify consent. The data collector will explain risks and benefits to potential enrollees before conducting the verbal autopsy and administering the household questionnaire in intervention and control clusters. Participants will be informed that they have the right to withdraw from the study at any time and that there are no penalties from doing this and this will not in any way affect their ability to receive any health care services.

   Ethical issues and Benefits The questionnaires will be designed to minimize the length of the interview, as the mother may be interviewed twice; at the follow up household visit on or after day 8 post-birth and in case of a verbal autopsy, thus, disrupting her routine.

   Culturally appropriate time interval (40 days) will be observed before approaching the family for a verbal autopsy in case of a stillbirth or perinatal death. The respondents will be able to skip any questions they are not comfortable with answering and stop the interview if they do not want to continue with it. The clinical audits and trainings will be conducted in such a way that the health care providers and community health workers do not feel vulnerable or persecuted in any way.

   Verbal Autopsy After the notification of a baby's death during the perinatal period, the data collector will make a home visit 40 days after the death. The parents will be given the choice of whether or not a verbal autopsy (Annex V) can be performed on the events surrounding the death of the newborns. If both parents are present, the verbal autopsy will be administered to the mother. If parents are not present, the data collector will ask if one of the parents will return home and be available for the interview within 24 hours. If a parent will not be available within 24 hours, the data collector will administer the verbal autopsy to an adult immediate relative who may be present (in order of priority: adult sibling to the deceased; grandparent; aunt or uncle to the deceased; cousin to the deceased). Consent will be obtained from whichever family member is the subject of the interview and if consent is obtained, they will be requested to answer the questions to the best of their personal knowledge. The data collector will explain that participation in the verbal autopsy is voluntary and that the respondent may choose to answer all, some, or no questions and may choose to stop the interview at any time without consequence. Observance of a 40 days grievance period between the death of a newborn and administration of the verbal autopsy will be mandatory for the data collectors due to local norms. The primary investigator and the co- primary investigator in this study have experience with the use of verbal autopsies associated with maternal, neonatal and child mortality related to obstetric causes. There are no known psychological or social risks associated with the verbal autopsy, additionally there is minimal potential for increased time-burden to the parents as a result of participating in the verbal autopsy. The verbal autopsy will be administered in the home of the respondent by a trained data collector and will take approximately 30-40 minutes to complete. Verbal autopsies will be administered in cases of perinatal deaths and stillbirths for newborns delivered in the CSComs and for newborns delivered at home but referred to a CSCom within the perinatal period. Each completed verbal autopsy will be independently reviewed by two local physicians and a cause of death will be assigned by them. If the two physicians do not assign the same diagnosis, a third physician (adjudicator) will review the two causes of death and assign a final cause of death.

ELIGIBILITY:
Inclusion Criteria:

* All CSComs providing basic obstetric care with at least one health care provider trained in AMTSL, ENC and PNC with data collection/ utilization in Koulikoro, Kolokani, Banamba and Dioïla study clusters.
* All community health workers reporting to an included CSCom.
* All CSCom deliveries (both mother and newborn) in study clusters and live home births referred to a facility within the perinatal period.
* Mother intending to maintain residence in study area for first week of newborn's life.

Exclusion Criteria:

* CSComs not providing basic obstetric care or not having trained maternal and neonatal health care providers in AMTSL, ENC and PNC and not collecting/utilizing data.
* CHW's will be excluded if linked to an in-eligible CSCom or if they have not been trained in the standard MoH CHW training curriculum.
* Failure to provide consent to enroll in study (intervention or control clusters).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Perinatal Mortality | First 7 days of life
  Deaths occurring within 7 days of birth and fetal deaths (stillbirth) per 1000 CSCOM births

SECONDARY OUTCOMES:
Resuscitation-Initiation of breathing | Immediately at birth
  Either the stimulation of the newborn, or the clearing of the airways using a suction bulb/catheter or using a bag and mask to resuscitate, per 1000 live births in a CSCOM.
Early initiation of breastfeeding | An hour after birth
  If child was breastfed within an hour of birth, per 1000 live births in a CSCOM.
Exclusive breastfeeding | First 7 days of life
  If child was given breastmilk and no other food or drink for the first 7 days of life, per 1000 live births in a CSCOM.
Thermal protection (dried and wrapped) | Immediately at birth
  If newborn was dried and wrapped immediately after birth, per 1000 live births in a CSCOM
Thermal protection (Kangaroo mother care) | Immediately at birth
  Immediately after birth was the newborn put on the chest of the mom - skin to skin, per 1000 live births in a CSCOM.
Clean cord care | First 7 days of life
  Newborns who had alcohol or chlorhexidine applied to the umbilical cord but nothing else, per 1000 live births in a CSCOM.
Delayed first bath | First 24 hours of life
  Newborn not bathed within first 24 hours of life, per 1000 live births in a CSCOM.
Newborn weighed | First 24 hours of life
  Newborn weight checked after birth, per 1000 CSCOM births.
Severe Infection | First 7 days of life
  Diagnosis of a severe infection, per 1000 CSCOM live births.
Neonatal hypothermia | First 7 days of life
  Diagnosis of neonatal hypothermia, per 1000 CSCOM live births.
Umbilical cord infection | First 7 days of life
  Diagnosis of umbilical cord infection per 1000 CSCOM live births.
Perinatal bleeding | First 7 days of life
  Diagnosis of perinatal bleeding per 1000 CSCOM live births
Postpartum hemorrhage | Immediately after delivery
  Postpartum hemorrhage of >= 500ml during childbirth in a CSCom, per 1000 deliveries
Obstructed labor - referral | During delivery
  # of women referred to a higher-level facility from a CSCOM due to obstructed labor, per 1000 deliveries.
Post-partum hemorrhage - referral | Immediately after delivery
  # of deliveries referred to a higher-level facility from a CSCOM due to post-partum hemorrhage, per 1000 deliveries.
Low birth weight - referral | First 7 days of life
  # of referrals for low birth weight from a CSCOM to a higher-level facility, per 1000 live births.
Moderate to severe hypothermia - referral | First 7 days of life
  # of referrals for moderate to severe hypothermia from a CSCOM to a higher level facility, per 1000 live births.
Severe infection - referral | First 7 days of life
  # of referrals for severe infection from a CSCOM to a higher level facility, per 1000 live births.
Moderate to severe umbilical cord infection - referral | First 7 days of life
  # of referrals for moderate to severe umbilical cord infection from a CSCOM to a higher level facility, per 1000 live births.

CONTACTS AND LOCATIONS:
Overall Officials: Diego G Bassani, Ph.D., Principal Investigator — The Hospital for Sick Children
Locations (1):
- iCCM Sites, Koulikoro, Mali

REFERENCES:
- [Derived] Zombre D, Kortenaar JL, Zareef F, Doumbia M, Doumbia S, Haidara F, McLaughlin K, Sow S, Bhutta ZA, Bassani DG. Combined Clinical Audits and Low-Dose, High-frequency, In-service Training of Health Care Providers and Community Health Workers to Improve Maternal and Newborn Health in Mali: Protocol for a Pragmatic Cluster Randomized Trial. JMIR Res Protoc. 2021 Dec 10;10(12):e28644. doi: 10.2196/28644. PMID 34889776